CLINICAL TRIAL: NCT00558467
Title: A Randomized, Double-blind, Placebo-controlled, Flexible Dose Study to Evaluate Efficacy and Safety of Pramipexole Immediate Release (0.125-0.5mg/Day) Versus Placebo for 6 Weeks in Children and Adolescents (Age 6-17 Inclusive) Diagnosed With Tourette Disorder According to DSM IV Criteria.
Brief Title: Pramipexole Pilot Phase II Study in Children and Adolescents With Tourette Disorder According to DSM-IV Criteria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.644
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-03

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pramipexole (Other)
  Interventions: Drug: pramipexole immediate release (IR)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pramipexole immediate release (IR)
  Arms: Pramipexole
Drug: Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, flexible dose study to evaluate efficacy and safety of Pramipexole versus placebo for 6 weeks in children (age 6-17) diagnosed with Tourette Disorder according to DSM IV criteria. The primary efficacy measure will be the Total Tic Score (TTS) of the Yale Global Tic Severity Scale (YGTSS) at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male of female patients 6-17 yrs.
* Written informed consent.
* Diagnosed with Tourette's Disorder with a > or equal to 22 on the Total Tic Score at baseline.
* Diagnosed with Tourette's Disorder when administering the Diagnostic Interview Schedule for Children.
* Having at least 1 tic/day.
* Women of childbearing age must have a negative serum pregnancy test at screening and must use a medically accepted contraceptive method.
* Either a newly diagnosed patient or a patient diagnosed with Tourette's Disorder who can safely discontinue treatment.
* Having a body weight of > or equal to 20 kg (44 lbs).

Exclusion Criteria:

* Any women of childbearing age having a positive serum pregnancy test at screening.
* Patients who have clinically significant renal disease or serum creatinine greater than 1.0 mg/dL at screening.
* Lab results at screening: hemoglobin below lower limit of normal which is determined to be clinically significant; Thyroid Stimulating Hormone (TSH), triiodothyronine (T3) or thyroxine (T4) clinically significant; clinically significant abnormalities in labs.
* Other clinically significant metabolic-endocrine, hematological, gastrointestinal disease, pulmonary disease which would preclude the patient from participating in this study.
* History of Schizophrenia or any psychotic disorder, history of mental disorders or any present Axis I psychiatric disorder according to Diagnostic and Statistic Manual of Mental Disorders Fourth Edition (DSM-IV) requiring any medical therapy except for patients with a diagnosis of attention deficit hyperactivity disorder (ADHD) or obsessive-compulsive disorder (OCD) who are not on therapy.
* History of/or clinical signs of epilepsy or seizures other than fever related seizures in early childhood.
* History of/or clinical signs of any malignant neoplasm.
* Allergic response to pramipexole.
* Had previous treatment with dopamine agonists other than pramipexole within 14 days prior to baseline visit.
* Had any other medical treatment for Tourette's Disorder besides the study medication within 28 days prior to baseline visit.
* Had withdrawal symptoms of any medication at screening or at the baseline visit.
* Having a Kaufman Brief Intelligence Test (KBIT IQ) score <70 at screening.
* Having a children's Yale-Brown obsessive-compulsive scale (CY-BOCS) score of >15 at baseline.
* Patients who meet criteria for Restless Legs Syndrome and or Periodic Limb Movement disorder.
* Patients with severe asthma.
* Patients that have initiated psychotherapy for Tourette's Disorder, OCD or ADHD within 3 mths of starting the trial.
* Patients receiving psychological, cognitive and/or behavioral treatments greater than 3 mths prior to start of trial for Tourette's Disorder, OCD, and/or ADHD who will have changes in treatment plan.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- United States (14):
  - 248.644.0026 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 248.644.0025 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 248.644.0006 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 248.644.0012 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.644.0005 Boehringer Ingelheim Investigational Site, Cambridge, Massachusetts
  - 248.644.0003 Boehringer Ingelheim Investigational Site, Manhasset, New York
  - 248.644.0009 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.644.0018 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.644.0013 Boehringer Ingelheim Investigational Site, Orangeburg, New York
  - 248.644.0029 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 248.644.0010 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 248.644.0030 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 248.644.0008 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 248.644.0023 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- Germany (2):
  - 248.644.49001 Boehringer Ingelheim Investigational Site, Hanover
  - 248.644.49004 Boehringer Ingelheim Investigational Site, Ulm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets matching the Pramipexole tablets to be taken per os
- Pramipexole: Pramipexole (tablets of 0.0625 mg, 0.125 mg and 0.25 mg) to be taken per os. Starting dose 0.0625 mg bid, with possible down titration after one week to 0.0625 mg qd or optional up titration to 0.125 mg bid, after the second week optional up titration to 0.125 mg tid, after the third week optional up titration to 0.25 mg bid.
Period: Overall Study
Arm/Group | Placebo | Pramipexole
Started | 20 | 43
Completed | 19 | 39
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Patient moving out of state | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pramipexole | Total
Number analyzed (Participants) | 20 | 43 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.1 (3.2) | 12.2 (2.4) | 11.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 18 | 35 | 53
Attention Deficit Hyperactive Disorder [Number; unit: Number of Patients] — Diagnosis of disorder was performed using National Institute of Mental Health Diagnostic Interview Schedule for Children (NIMH DISC IV) and resulted in patients being classified as negative diagnosis, intermediate diagnosis and positive diagnosis for disorder.
  Number of Patients
    Intermediate | 3 | 6 | 9
    Negative | 9 | 22 | 31
    Positive | 8 | 15 | 23
Duration of Tourettes syndrome [Number; unit: participants]
  1-5 years | 10 | 19 | 29
  Less than 1 years | 6 | 12 | 18
  More than 5 years | 4 | 12 | 16
Ethnicity, Customized [Number; unit: Number of Patients]
  Hispanic/Latino | 2 | 5 | 7
  Not Hispanic/Latino | 18 | 38 | 56
Obsessive Compulsive Disorder [Number; unit: participants] — Diagnosis of disorder was performed using National Institute of Mental Health Diagnostic Interview Schedule for Children (NIMH DISC IV) and resulted in patients being classified as negative, intermediate and positive for disorder.
  participants
    Intermediate | 1 | 3 | 4
    Negative | 16 | 37 | 53
    Positive | 3 | 3 | 6
Race, Customized [Number; unit: participants]
  Black/African American | 2 | 4 | 6
  White | 18 | 39 | 57
Body Mass Index [Mean (Standard Deviation); unit: kilograms/(meters squared)] | 20.085 (5.324) | 22.575 (5.656) | 21.784 (5.632)
Height [Mean (Standard Deviation); unit: centimeters] | 150.7 (21.6) | 155.3 (16.2) | 153.8 (18)
Weight [Mean (Standard Deviation); unit: kilograms] | 47.48 (21.29) | 55.87 (20.64) | 53.21 (21.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Tic Score of the Yale Global Tic Severity Scale
Description: Total Tic Score is the sum of ten individual ratings of the impairment due to tics. Each scale ranges from 0 (None/Absent) to 5 (Severe) and total score ranges from 0 to 50.
  Analysis was adjusted for baseline total tic score and age as linear covariates.
Time Frame: baseline 6 weeks
Population: The Full Analysis Set (FAS) with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
score on a scale | -7.17 (2.02) | -7.16 (1.38)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.996, ANCOVA; Least Squares mean difference = 0.01, 95% CI 2-sided [-4.95 to 4.97]

2. Secondary Outcome: Mean Change From Baseline in Total Tic Score of the Yale Global Tic Severity Scale at Week 1
Description: Total Tic Score is the sum of ten individual ratings of the impairment due to tics. Each scale ranges from 0 (None/Absent) to 5 (Severe) and total score ranges from 0 to 50
Time Frame: baseline 1 week
Population: The Full Analysis Set was composed of patients that provided a baseline and a post-baseline assessment in Total Tic Score. A total of 62 patients are included in the Full Analysis Set, 20 placebo patients and 42 pramipexole patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
score on a scale | -3.7 (4.1) | -4.1 (5.4)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; Repeated Measures; Least square means difference = -3.94, 95% CI 2-sided [-5.81 to -2.08]

3. Secondary Outcome: Mean Change From Baseline in Total Tic Score of the Yale Global Tic Severity Scale at Week 2
Description: as for outcome 2
Time Frame: baseline and 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 41
score on a scale | -5.3 (7.9) | -5 (7.4)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; Repeated measures; Least square means difference = -5.30, 95% CI 2-sided [-7.21 to -3.39]

4. Secondary Outcome: Mean Change From Baseline in Total Tic Score of the Yale Global Tic Severity Scale at Week 3
Description: as for outcome 2
Time Frame: baseline and 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 41
score on a scale | -6.2 (6.3) | -5.4 (6.3)

5. Secondary Outcome: Mean Change From Baseline in Total Tic Score of the Yale Global Tic Severity Scale at Week 4
Description: as for outcome 2
Time Frame: baseline and 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 40
score on a scale | -6 (7.9) | -6.4 (7.3)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; Repeated measures; Least square means difference = -5.97, 95% CI 2-sided [-7.88 to -4.06]

6. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale Due to Motor and Phonic Tics at Week 6
Description: Total Score is a rating of the overall impairment due to motor and phonic tics. The scale ranges from 0 (None) to 50 (Severe)
Time Frame: baseline and 6 weeks
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
score on a scale | -15.43 (4.44) | -15.58 (3.03)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.9780, ANCOVA; Least Squares Mean differnce = -0.15, 95% CI 2-sided [-11.05 to 10.75]

7. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale Due to Motor and Phonic Tics at Week 1
Description: as for outcome 6
Time Frame: baseline 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
score on a scale | -6.2 (13.3) | -8.8 (11.1)

8. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale Due to Motor and Phonic Tics at Week 2
Description: as for outcome 6
Time Frame: baseline and 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 41
score on a scale | -9.5 (16.1) | -10.6 (17.5)

9. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale Due to Motor and Phonic Tics at Week 3
Description: as for outcome 6
Time Frame: baseline and 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 41
score on a scale | -14.1 (17.2) | -12.2 (15.7)

10. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale Due to Motor and Phonic Tics at Week 4
Description: as for outcome 6
Time Frame: baseline 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 40
score on a scale | -15.5 (18.2) | -13.9 (15.7)

11. Secondary Outcome: Clinical Global Impressions - Improvement at 1 Week
Description: Overall improvement during the last week compared to baseline ranging from 1 (very much improved), 2 (much improved), to 7 (very much worse). Responder has 'very much' or 'much' improvement. Non responder has less improvement than 'much' improvement.
Time Frame: baseline and Week 1
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 0 | 5
  Not Responder | 20 | 37
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.1052, Cochran-Mantel-Haenszel

12. Secondary Outcome: Clinical Global Impressions - Improvement at Week 2
Description: as for outcome 11
Time Frame: baseline and Week 2
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 1 | 6
  Not Responder | 19 | 36
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.2274, Cochran-Mantel-Haenszel

13. Secondary Outcome: Clinical Global Impressions - Improvement at Week 3
Description: as for outcome 11
Time Frame: baseline and Week 3
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 2 | 5
  Not Responder | 18 | 37
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.7691, Cochran-Mantel-Haenszel

14. Secondary Outcome: Clinical Global Impressions - Improvement at Week 4
Description: as for outcome 11
Time Frame: baseline and Week 4
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 7 | 6
  Not Responder | 13 | 36
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0674, Cochran-Mantel-Haenszel

15. Secondary Outcome: Clinical Global Impressions - Improvement at Week 6
Description: as for outcome 11
Time Frame: baseline and Week 6
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 7 | 11
  Not Responder | 13 | 31
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.4944, Cochran-Mantel-Haenszel

16. Secondary Outcome: Clinical Global Impressions - Severity of Illness at Week 1
Description: Assessment of the overall severity of illness on a scale ranging from 1 (not at all ill) to 7 (the most extremely ill patients). Improved, Unchanged and Worsened responses correspond to changes from baseline of: -2 or less, -1 to +1, and 2 or greater.
Time Frame: baseline and Week 1
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Improved | 0 | 4
  Unchanged | 20 | 38
  Worsened | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.162, Cochran-Mantel-Haenszel

17. Secondary Outcome: Clinical Global Impressions - Severity of Illness at Week 2
Description: as for outcome 16
Time Frame: baseline and Week 2
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Improved | 1 | 4
  Unchanged | 19 | 37
  Worsened | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.6375, Cochran-Mantel-Haenszel

18. Secondary Outcome: Clinical Global Impressions - Severity of Illness at Week 3
Description: as for outcome 16
Time Frame: baseline and Week 3
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Improved | 3 | 4
  Unchanged | 17 | 37
  Worsened | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.6625, Cochran-Mantel-Haenszel

19. Secondary Outcome: Clinical Global Impressions - Severity of Illness at Week 4
Description: as for outcome 16
Time Frame: baseline and Week 4
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Improved | 4 | 4
  Unchanged | 16 | 38
  Worsened | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.2664, Cochran-Mantel-Haenszel

20. Secondary Outcome: Clinical Global Impressions - Severity of Illness at Week 6
Description: as for outcome 16
Time Frame: baseline and Week 6
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Improved | 4 | 10
  Unchanged | 16 | 32
  Worsened | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.7302, Cochran-Mantel-Haenszel

21. Secondary Outcome: Patient Global Impression at Week 1
Description: Assessment of the change of the patient's overall condition during the last week compared to the patient's condition at baseline on a scale ranging from 1 (very much better) to 7 (very much worse). A responder is defined as having a response of very much (1) or much better (2).
Time Frame: baseline and Week 1
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 4 | 7
  Not Responder | 16 | 35
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.7723, Cochran-Mantel-Haenszel

22. Secondary Outcome: Patient Global Impression at Week 2
Description: as for outcome 21
Time Frame: baseline and Week 2
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 6 | 9
  Not Responder | 14 | 33
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.4852, Cochran-Mantel-Haenszel

23. Secondary Outcome: Patient Global Impression at Week 3
Description: as for outcome 21
Time Frame: baseline and Week 3
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 5 | 7
  Not Responder | 15 | 35
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.4607, Cochran-Mantel-Haenszel

24. Secondary Outcome: Patient Global Impression at Week 4
Description: as for outcome 21
Time Frame: baseline and Week 4
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 4 | 7
  Not Responder | 16 | 35
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.7723, Cochran-Mantel-Haenszel

25. Secondary Outcome: Patient Global Impression at Week 6
Description: as for outcome 21
Time Frame: baseline and Week 6
Population: The Full Analysis Set with last observation carried forward (LOCF).
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 20 | 42
Number of Patients
  Responder | 6 | 12
  Not Responder | 14 | 30
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.9389, Cochran-Mantel-Haenszel

26. Secondary Outcome: Clinically Significant Abnormalities in Vital Signs (Orthostatic Reaction and Pulse Rate), and Serum Chemistry.
Time Frame: baseline and Week 6
Population: Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 19 | 40
participants
  Phosphate - increase | 2 | 5
  Bilirubin, total - increase | 0 | 1
  Tachycardia | 0 | 1
  Orthostatic hypotension | 1 | 4

ADVERSE EVENTS:
Time Frame: All events with an onset after the first dose of study medication and up to a period of 48 hours after the last dose of study medication were assigned to the treatment period.
Arm/Group | Placebo | Pramipexole
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/43
Other Adverse Events (participants affected / at risk) | 13/20 | 25/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Pramipexole (N=43)
Gastroenteritis viral (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Pramipexole (N=43)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 0 | 5
Fatigue (General disorders) | 2 | 4
Pyrexia (General disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 5 | 12
Somnolence (Nervous system disorders) | 1 | 3
Sleep disorder (Psychiatric disorders) | 0 | 3
Tic (Psychiatric disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.